CLINICAL TRIAL: NCT06214585
Title: Effect of Intermittent Heat & Cold Versus Heat Only Therapy on Comfort and Duration of Labor Among Primigravida
Brief Title: Effect of Intermittent Heat and Cold Therapy on Comfort During Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University, Nepal (Other)
Responsible Party: Principal Investigator, Isabel Lawot, Lecturer, Tribhuvan University, Nepal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ShardaU
Record Dates: First submitted 2023-12-14; First posted 2024-01-19 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Labour Pain; Cold Therapy; Heat Therapy
Keywords: Comfort, Cold , Heat Therapy, Labor Pain
MeSH Terms: conditions — Labor Pain; Hyperthermia; Common Cold

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent Heat & cold Therapy (Experimental): There will be one group that will be receiving warm water application on the mother's back and then receiving ice pack application on the same region.
  Interventions: Procedure: Intermittent heat and cold versus heat-only therapy; Procedure: Heat- only Therapy
- Heat- Only Therapy (Experimental): This group of mothers will receive a warm application by hot water bag only on her back
  Interventions: Procedure: Intermittent heat and cold versus heat-only therapy; Procedure: Heat- only Therapy
- Control Group (No Intervention): This group will receive just standard care as hospital protocol

INTERVENTIONS:
Procedure: Intermittent heat and cold versus heat-only therapy — for the experimental group, a cyclical method of alternating heat and cold application will be used on the lumbosacral and lower abdominal area of the laboring women. The process involves applying a hot pack with a temperature range of 38-40°C on their lower abdomen and low back for 30 minutes during contractions and a relaxing period using a 2-litre rubber hot water bag. Subsequently, reusable ice packs typically contain water, covered with a towel and with a temperature range of 0-5°C will be applied to the same areas for 10 minutes. After a 30-minute interval, the heat application will be reapplied, and this alternating heat and cold cycle will be repeated throughout the first stage of the laboring process.
  Arms: Heat- Only Therapy; Intermittent Heat & cold Therapy
Procedure: Heat- only Therapy — hot water bag will be used to provide heat to the lower back of primigravida women during the first stage of labor. The water in the bag will be maintained at a temperature of 40-42ºC. The application of heat will last for 20 minutes, and it will be repeated every hour until the cervix is fully dilated.
  Arms: Heat- Only Therapy; Intermittent Heat & cold Therapy

SUMMARY:
Summary of the Study Childbirth is one of the most significant and complex experiences in any mother's life. According to a study, labour pain ranges from mild to severe and is felt throughout the body, particularly in the lower abdomen, vagina, and around the waist. The mean pain perception of the prurient as assessed by the Visual Analog scale (VAS) was 7.0 with a range of 1.2-10.0. In a study, 50% of parturients rated labour pain as severe (VAS > 7.1). The majority of the respondents 86.4% desired some form of pain relief. Pain relief during labor is a crucial component of the labor process. Non-drug techniques for alleviating labor pain focus on psychological and physical discomfort elements. A study in Panjab was performed to assess the effectiveness of heat therapy on the lower back among women in labor pain during the first stage of labor and found that heat therapy reduces the severity of pain in the first stage of labor. A study performed in India found that intermittent heat and cold therapy successfully shorten the first and second stages of labor's duration and pain. The purpose of the study is to compare the impact of intermittent heat and cold therapy with heat-only therapy on comfort and duration of labor among primigravida women at a Bharatpur hospital in Nepal.

A quantitative research approach will be adopted and the research design will be a true experimental pretest posttest design. It will be conducted among 150 low-risk primigravida women aged 20 to 35 years with a gestation of 37-41 weeks of pregnancy admitted to the maternity of Bharatpur Hospital, Chitwan Nepal who are anticipated to deliver spontaneously. The participants will be divided into 50 in each 3 groups. One group will receive intermittent heat and cold therapy, another group will receive heat-only therapy and one group will be the control group. The tool will be a standard tool which are Visual Analog Scale (VAS) and Childbirth Comfort Questionnaire (CCQ). All the ethical clearance will be obtained before collecting data from Sharda University, Nepal Health Research Council, and Bharatpur Hospital. Informed consent will be taken from all the participants and their rights, privacy, confidentiality, and comfort will be maintained. The participants can withdraw from the study at any time without giving any explanation. The data will be organized and entered into Statistical Package of Social Sciences (SPSS) version 16 for analysis. The data will be analyzed according to the objectives of the study by using descriptive and inferential statistics.

DETAILED DESCRIPTION:
Heat Only Therapy A 2-liter rubber hot water bag will be utilized to provide heat to the lower back of primigravida women during the first stage of labor. The water in the bag will be maintained at a temperature of 40-42ºC. The application of heat will last for 20 minutes, and it will be repeated every hour until the cervix is fully dilated. To prepare the hot water, tap water will be boiled in a stainless steel pot until it reaches 70ºC. Before filling the hot water bag, its temperature will be verified using a laboratory thermometer. The bag will then be covered with a towel and applied to the laboring women, ensuring the heat is tolerable for her. If the temperature falls below the specified range, another hot water bag will be made ready for replacement. Intermittent Heat & Cold Therapy During the first stage of labor (from 4-5 to 10 cm of cervical dilation) for the experimental group, a cyclical method of alternating heat and cold application will be used on the lumbosacral and lower abdominal area of the laboring women. The process involves applying a hot pack with a temperature range of 38-40°C on their lower abdomen and low back for 30 minutes during contractions and a relaxing period using a 2-litre rubber hot water bag.

Subsequently, reusable ice packs typically contain water, covered with a towel and with a temperature range of 0-5°C will be applied to the same areas for 10 minutes. After a 30-minute interval, the heat application will be reapplied, and this alternating heat and cold cycle will be repeated throughout the first stage of the laboring process. After interventions 4-5, 7-8 and 9-10 cm of cervical dilation, we will assess the comfort including pain level and after 10 cm of cervical dilation, duration will be calculated to identify the total duration of first stage of labor

ELIGIBILITY:
Inclusion Criteria:

Low-risk primigravida are those pregnant women who are between the ages of 18 to 35 years old admitted to Bhartpur hospitals and anticipated normal delivery.

* Completed 4 ANC visits
* Normal size fetus and without any complication by USG scan
* Weeks of gestation 37 to 41
* No history of abortions
* Who had not taken any analgesic and other regular medication
* Normal BMI (Pre-pregnancy 18.5-24.9)
* Women willing to participate
* Those mothers who are initial phase of labor

Exclusion criteria ('no any complication')

* Pregnant women who had a history of abortion
* Pregnancy-induced hypertension and heart conditions(pre/eclampsia)
* Antepartum haemorrhage
* Pregnancy with urinary system disease such as UTI
* Hyper or hypothyroidism
* Anemia
* Obesity
* Pregnancy with Diabetes
* Diagnosed Mental Illnesses such as Stress anxiety depression, Psychosis or epilepsy
* Any Physical Disability
* Fever during Labor
* Those pregnant women who did not have any antenatal visit
* Pregnant women who will not willing to participate
* Those women who develop complications during the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Level of Comfort | 1 to 2 hours of intervention
  It will be measured using Childbirth Comfort Questionnaire.The Childbirth Comfort Questionnaire (CCQ) was developed and tested in 2002-2003. Face validity was accomplished by a panel of experts: midwives, obstetricians, labor and delivery nurses and women who had given birth. The instrument has a 0.71 Cronbach's (sample size n = 64). The instrument is administered twice during labor: latent & active phase. To score, reverse code the negative responses and total the sum. Higher totals mean higher comfort.
Duration of Labor | 4 to 5 hours
  Duration of labor will be measured using a partograph. The initiation of labor time to completion labor process will be recorded in the partograph. At the end of the first labour stage, the total labour hour will be caculated and mentioned as mean duration which will be compared with other data
Level of labor pain | 1 to 2 hours of intervention
  A Visual Analogue Scale will be used as the pain rating scale used for the first time in 1921 by Hayes and Patterson. There is no pain" on the far left and "the most intense pain imaginable" on the far right. In between these two extremes, words such as mild, moderate, severe, and very severe pain are assigned to each 2 cm distance on the line, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Bharatpur Hospital, Bharatpur, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Undecided